CLINICAL TRIAL: NCT01584921
Title: Renal Effects of Erythropoietin in Humans
Acronym: EPO 2012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Niels Jacob Aachmann-Andersen, Medical doctor, phd.-student, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-2-2011-068
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Renal Effects
Keywords: Erythropoietin; Glomerular filtration rate; Tubular reabsorption; Renal function; Renal perfusion
MeSH Terms: interventions — Erythropoietin; epoetin beta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 1 ml of saline (Sodium Chloride 9 mg/ml) is given subcutaneously before 10 O-clock a.m. on day 1,2,3,5,7,9,11 and 13. On day 1,2 and 3 six ml in total is given in six syringes in order to maintain the double blinding.
  Interventions: Drug: Placebo
- Low dose Erythropoietin (Active Comparator)
  Interventions: Drug: Erythropoietin (Epoetin-beta, NeoRecormon®)
- High dose Eryhropoietin (Active Comparator)
  Interventions: Drug: Erythropoietin (Epoetin-beta, NeoRecormon®)

INTERVENTIONS:
Drug: Erythropoietin (Epoetin-beta, NeoRecormon®) — 5000 IU/ml of NeoRecormon (Epoetin beta) is given subcutaneously as one ml before 10 O-clock a.m. on day 1,3,5,7,9,11 and 13. On day 1 and 3 5000 IU is given in one syringe and five ml of saline in total is given in five other syringes in order to maintain the double blinding. On day 2 six syringes of a total of 6 ml of saline is given in six syringes.
  Arms: Low dose Erythropoietin
Drug: Erythropoietin (Epoetin-beta, NeoRecormon®) — 30.000 IU of NeoRecormon (Epoetin beta) is given subcutaneously as a total of six ml (5.000 IU/ml) given in six syringes before 10 O-clock a.m. on day 1,2 and 3.
  On day 5,7,9,11 and 13 six ml of saline in total is given in six syringes in order to maintain the double blinding.
  Arms: High dose Eryhropoietin
Drug: Placebo — 1 ml of saline (Sodium Chloride 9 mg/ml) is given subcutaneously before 10 O-clock a.m. on day 1,2,3,5,7,9,11 and 13. On day 1,2 and 3 six ml in total is given in six syringes in order to maintain the double blinding.
  Arms: Placebo

SUMMARY:
Erythropoietin (EPO) is a glycoprotein produced mainly in the kidney. After its release to the bloodstream EPO binds to its receptor predominantly located within the bone marrow where erythropoiesis is stimulated. Recently, we have shown that recombinant human EPO (rHuEPO) down-regulates circulating levels of renin and aldosterone. Concomitant clearance studies revealed a decrease in proximal tubular reabsorption of sodium and water and a fall in glomerular filtration rate (GFR). These results for the first time demonstrate a link between EPO and renal function: By inhibiting proximal tubular reabsorption, which in turn results in rapid declines in GFR and renin/aldosterone levels, EPO may directly reduce the major oxygen consuming factor in the kidney. The expected result will be an increase of the oxygen tension in the environment of renal EPO producing cells, in this way initiating an appropriate signal for down-regulation of endogenous EPO synthesis when circulating levels of EPO are high.

The aim of this project is to test this hypothesis by investigating the renal effects of rHuEPO in humans. In a double-blinded manner healthy subjects will be tested with placebo, or low-dose rHuEPO for two weeks, or high-dose rHuEPO for three days. Accurate sodium balance studies will be conducted together with renal clearance studies for measurements of renal plasma flow (131I-Hippuran clearance with renal venous sampling), GFR (51Cr-EDTA clearance) and the segmentel tubular handling of sodium and water (lithium clearance).

EPO is the sole haematopoietic growth factor that is mainly produced in the kidneys and the project will provide new information about basic physiological issues regarding the association between renal function and the regulation of EPO synthesis.

DETAILED DESCRIPTION:
The haematopoietic effect of EPO and rHuEPO has been known for five decades but still the exact mechanisms for regulation of EPO synthesis in the kidneys remain unclear. Recently, we confirmed our previous observation that rHuEPO in normal subjects produces arterial hypertension and a reduction in plasma volume. Moreover, the study delineated the time course of these changes: rHuEPO promptly, and before any changes in hematocrit, blood volumes and blood pressure can be detected, causes a down-regulation of the renin-aldosterone system, proximal tubular reabsorption and GFR.

The effect of rHuEPO on arterial blood pressure has been demonstrated to occur independent of its haematopoietic effect and subsequent effect on blood viscosity. Recently, we reported that also short-time administration of very high doses of rHuEPO (30,000 IU/day for three days) increases arterial blood pressure and the blood pressure response to exercise to a similar extent as prolonged, low-dose rHuEPO for three month. The exact mechanisms remains unclear, but may involve rHuEPO induced release of endothelin and inhibition of eNOS mediated production of NO.

The early rHuEPO induced reduction of renin and aldosterone was not caused by changes in plasma and blood volumes. A fall in intravascular volume normally leads to the opposite effect due to a decreased NaCl load to the macula densa and an increased sympathetic stimulation of the juxtaglomerular apparatus. The link between administration of rHuEPO and the renin-angiotensinaldosterone system is interesting because the production of endogenous EPO is regulated by this system. Administration of angiotensin II in humans stimulates EPO synthesis and, conversely, inhibitors of angiotensin converting enzyme and angiotensin II receptors decrease the plasma concentration of endogenous EPO. In patients with type-1 diabetes, an inherent high activity of basal renin-angiotensin system (in part governed by genetic factors) was associated with higher levels of EPO compared to patients with a low activity of basal renin-angiotensin system. Our results suggest that rHuEPO may activate an opposite pathway so as to down-regulate the activity of the renin-angiotensin-aldosterone system independent of changes in red blood cell mass, blood volumes and blood pressure.

Our renal clearance data suggest that the rHuEPO-induced inhibition of the renin-aldosterone system is associated with a reduction of absolute proximal tubular reabsorption of fluid and a fall in GFR. Changes in end-proximal delivery of tubular fluid to the macula densa produce inverse changes in renin release and thus the suppression of plasma renin levels may be secondary to direct effects of rHuEPO on proximal tubular reabsorption. In addition, a decrease in proximal tubular reabsorption activates the tubuloglomerular feedback mechanism causing a parallel decrease in GFR. The exact molecular mechanisms for rHuEPO's effect on the proximal tubule remain unknown but may involve inhanced release of renal endothelin-1 which in low doses attenuates sodium reabsorption in the proximal tubule. Tubular reabsorption of sodium is the main oxygen consuming process in the kidney and around 70 % of the filtered load is reabsorbed in the proximal tubule. By inhibiting proximal tubular reabsorption, which in turn results in rapid declines in GFR and renin/aldosterone levels, rHuEPO may directly reduce the major oxygen consuming factor in the kidney, reduce the filtered load, and decrease angiotensin II and aldosterone dependent reabsorption in more distal nephron segments. Thus, we suggest that the renal effects of rHuEPO may be part of a feedback system that serves to down-regulate the endogenous renal synthesis of EPO in the presence of high levels of circulating EPO. In support of such a feedback system, evidence exists to indicate that prolonged administration of rHuEPO results in a suppression of urinary excretion of endogenous EPO, and also the renal effects of rHuEPO fits well in the hypothesis advanced by Donnelly, arguing that the kidney operates as a 'critmeter' to regulate the EPO synthesis and body haematocrit through the metabolic signal of renal tissue oxygen pressure.

It has been suggested that the reduction in plasma volume induced by rHuEPO may be caused by the hyporeninemic hypoaldosteronism leading to natriuresis. In our previous study we did not perform actual sodium balance studies. However, the renal sodium loss necessary to account for the observed decrease in plasma volume is small, and it is possible that the net effect of rHuEPO was to cause a negative sodium balance during the entire 28 days treatment period.

Hypotheses

1. rHuEPO decreases renal proximal tubular reabsorption, concentrations of renin and aldosterone, GFR, and overall renal perfusion.
2. In subjects on a sodium-fixed diet, rHuEPO increases the sodium excretion causing a negative sodium balance.
3. rHuEPO decreases renal oxygen consumption so as to augment oxygen tension at EPOproducing, interstitiel fibroblast-like cells in the juxtamedullary region.
4. rHuEPO decreases renal synthesis and secretion of endogenous EPO.
5. Blockade with specific endothelin antagonists (Bosantan) inhibits the renal effects of rHuEPO.

Research plan and methods The project includes normal subjects in which rHuEPO is administered according to previous protocols used by our group. In separate series subjects are given either 1) placebo, 2) rHuEPO (5,000 IU) every second day in two weeks, 3) rHuEPO (30,000 IU/day) for three days. Measurements are obtained at days 4, 11, 28. The trials are planned to be conducted in a double-blinded, cross-over design by which the subjects are randomised to three consecutive trial periods with either placebo, low-dose rHuEPO or high-dose rHuEPO separated by at least six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 20-40 years
* Non smoker for min. a year
* BP below 140/90
* No medicine use
* BMI below 25

Exclusion Criteria:

* Participation in other medical trails
* Allergi towards Erythropoietin
* Malignity diseases
* Epilepsy
* Staying above 1500 meters within the last 3 months
* Polycythemia
* Elite athlete
* Haematocrit above 55%

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in the Renal Blood Flow (RBF ml/min). | Day 4 and 25
  Renal clearance studies with timed urine collections and renal venous catherization for measurements of renal perfusion (131I-Hippuran).

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR ml/min) | Day 4, 11 and 25
  Renal clearance studies with timed urine collections for measurements of GFR (51Cr-EDTA) and segmental renal handling of sodium and water (lithium clearance).
Segmental renal handling of sodium and water (lithium clearance). | Day 4, 11 and 25.
  Renal clearance studies with timed urine collections and measurements of segmental renal handling of sodium and water (lithium clearance). All subjects will be studied during a sodiumfixed diet, with Lithiumcarbonat 300 mg given the evening before each studyday.
Blood and plasma volume | Day 4, 11 and 25
  With CO method blood and plasma volume are measured.
Analysis of hormones and proteins. | Day 4, 11 and 25.
  Analysis of concentrations of rHuEPO, EPO, renin, aldosterone, endothelin-1, nitrite/nitrate, citrulline, sodium and asymmetric dimethylarginine in urine, renal venous blood and venous blood.
Endothel function | Day 4, 11 and 25
  Endothel function measured with non-invasive arteriel tonometri (Endopat 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Niels Vidiendal Olsen, M.D., D.M.Sc., Study Chair — Department of Neuroscience and Pharmacology, University of Copenhagen
Locations (1):
- Department of Clinical Physiology and Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Copenhagen East, Denmark

REFERENCES:
- [Background] Olsen NV, Aachmann-Andersen NJ, Oturai P, Munch-Andersen T, Borno A, Hulston C, Holstein-Rathlou NH, Robach P, Lundby C. Erythropoietin down-regulates proximal renal tubular reabsorption and causes a fall in glomerular filtration rate in humans. J Physiol. 2011 Mar 15;589(Pt 6):1273-81. doi: 10.1113/jphysiol.2010.194241. Epub 2010 Aug 19. PMID 20724370
- [Background] Lundby C, Olsen NV. Effects of recombinant human erythropoietin in normal humans. J Physiol. 2011 Mar 15;589(Pt 6):1265-71. doi: 10.1113/jphysiol.2010.195917. Epub 2010 Aug 31. PMID 20807784
- [Background] Holstein-Rathlou NH. A closed-loop analysis of the tubuloglomerular feedback mechanism. Am J Physiol. 1991 Nov;261(5 Pt 2):F880-9. doi: 10.1152/ajprenal.1991.261.5.F880. PMID 1951720
- [Background] Jelkmann W. Erythropoietin: structure, control of production, and function. Physiol Rev. 1992 Apr;72(2):449-89. doi: 10.1152/physrev.1992.72.2.449. No abstract available. PMID 1557429
- [Background] Hutchings M, Hesse B, Gronvall J, Olsen NV. Renal 131I-hippuran extraction in man: effects of dopamine. Br J Clin Pharmacol. 2002 Dec;54(6):675-7. doi: 10.1046/j.1365-2125.2002.t01-5-01689.x. PMID 12492618
- [Background] Krapf R, Hulter HN. Arterial hypertension induced by erythropoietin and erythropoiesis-stimulating agents (ESA). Clin J Am Soc Nephrol. 2009 Feb;4(2):470-80. doi: 10.2215/CJN.05040908. PMID 19218474
- [Background] Rasmussen P, Foged EM, Krogh-Madsen R, Nielsen J, Nielsen TR, Olsen NV, Petersen NC, Sorensen TA, Secher NH, Lundby C. Effects of erythropoietin administration on cerebral metabolism and exercise capacity in men. J Appl Physiol (1985). 2010 Aug;109(2):476-83. doi: 10.1152/japplphysiol.00234.2010. Epub 2010 Jun 3. PMID 20522733
- [Background] Kristensen PL, Hoi-Hansen T, Olsen NV, Pedersen-Bjergaard U, Thorsteinsson B. Erythropoietin during hypoglycaemia in type 1 diabetes: relation to basal renin-angiotensin system activity and cognitive function. Diabetes Res Clin Pract. 2009 Jul;85(1):75-84. doi: 10.1016/j.diabres.2009.01.008. Epub 2009 Feb 10. PMID 19211168